CLINICAL TRIAL: NCT01834144
Title: The VIGORous Physical Activity for Glycaemic Control in Type 1 Diabetes (VIGOR) Trial
Acronym: VIGOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for the study was not renewed
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Institute of Child Health (Industry)
Responsible Party: Principal Investigator, Jon McGavock, Associate Professor, Dept. Of Pediatrics and Child Health, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B2012:136
Record Dates: First submitted 2013-03-27; First posted 2013-04-17 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Hypoglycaemia; Glycaemic variability; Vigorous Intensity Physical Activity; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate intensity exercise (Active Comparator): 150-200 minutes of weekly moderate intensity exercise (45-55% of peak fitness)
  Interventions: Other: Exercise Training
- Moderate + Vigorous Intensity Exercise (Active Comparator): 150-200 minutes of weekly moderate intensity exercise, with short bouts of vigorous intensity exercise (80-90% of peak fitness)
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training

SUMMARY:
Background/Justification: Regular physical activity (PA) has substantial health benefits in persons with type 1 diabetes (T1D), including reduced risk of complications and cardiovascular mortality. Despite these benefits, individuals with T1D remain significantly less active than their peers without diabetes. Two major factors likely explain the low rates of PA in young people with T1D: (1) fear of post-exercise hypoglycaemia, particularly nocturnal hypoglycaemia, and (2) a lack of empirical evidence for the efficacy of PA for achieving optimal glycaemic control. A number of acute exercise trials recently demonstrated that the inclusion of vigorous intensity PA in conventional moderate intensity (i.e. walking) PA sessions may overcome these limitations. No studies have tested the efficacy of high intensity PA for reducing the risk of exercise-related hypoglycaemia or glycaemic variability in a randomized controlled trial (RCT).

Study Hypotheses: In persons 15-35 years of age living with T1D, this study will test the hypotheses that (1) the addition of intermittent vigorous intensity PA to a moderate intensity intervention will reduce the time spent in hypoglycaemia in the 12 hour period following exercise and (2) the addition of intermittent vigorous intensity PA to a moderate intensity PA intervention will elicit significant improvements in glycemic excursions, as measured by the Mean Amplitude of Glycaemic Excursions (MAGE), in the 12-hour period following exercise.We are also exploring the hypothesis that reducing the risk of hypoglycemia will lead to a sustained increase in physical activity one year after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age: 15-45 years old
* Have lived with type 1 diabetes for at least 2 years
* HbA1c <9.9%
* Currently physically inactive (<150 minutes of self-reported structured physical activity per week)
* Undergone a resting ECG to screen for left ventricular hypertrophy, arrhythmias or signs or coronary artery disease that may be exacerbated with vigorous intensity exercise

Exclusion Criteria:

* Have frequent and unpredictable hypoglycaemia
* Had a change in insulin management strategy, including adoption of a pump, within 2 months of enrolment
* Are currently participating in structured activity or sport-related activities
* Are women who are pregnant or planning to get pregnant within the 12 months of the trial and those who are breastfeeding
* Have conditions that would render physical activity contraindicated including: uncontrolled hypertension (BP>150mmHg systolic or >95mmHg diastolic in a sitting position); severe peripheral neuropathy; history of cardiovascular disease
* Have a cognitive deficit resulting in an inability to provide informed consent
* Currently taking beta blockers
* Currently taking atypical antipsychotics or corticosteroids

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06-15 (Actual); Study Completion 2015-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Manitoba Institute of Child Health, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - University of Ottawa, Ottawa, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Intensity Exercise: 150-200 minutes of weekly moderate intensity exercise (45-55% of peak fitness)
  Exercise Training
- Moderate + Vigorous Intensity Exercise: 150-200 minutes of weekly moderate intensity exercise, with short bouts of vigorous intensity exercise (80-90% of peak fitness)
  Exercise Training
Period: Overall Study
Arm/Group | Moderate Intensity Exercise | Moderate + Vigorous Intensity Exercise
Started | 1 | 3
Completed | 1 | 2
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Intensity Exercise | Moderate + Vigorous Intensity Exercise | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 0 (0) | 0 (0) | 0 (0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Study funding not renewed; do data analyzed
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Hypoglycaemia in the 12-hour Period Following Exercise, Defined as an Interstitial Glucose Reading <4.0mmol/L and Measured by Continuous Glucose Monitor.
Time Frame: Measured at baseline, and 1, 8,16 and 52 weeks following randomization
Arm/Group | Moderate Intensity Exercise | Moderate + Vigorous Intensity Exercise
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Glycaemic Variability, Measured by the Mean Amplitude of Glycaemic Excursions (MAGE), in the 12-hour Period Following Exercise. This is Calculated From the Same Continuous Glucose Monitor Data as the Primary Outcome.
Time Frame: Measured at baseline, and 1, 8, 16 and 52 weeks following randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Moderate Intensity Exercise | Moderate + Vigorous Intensity Exercise
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No